CLINICAL TRIAL: NCT06016010
Title: Efficacy and Safety of USL for Dry Eye Disease (DED): a Randomized, Double-blind, Placebo-controlled, Parallel, Phase 2 Clinical Trial
Brief Title: Efficacy and Safety of USL for Dry Eye Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chan-Sik Kim (Other Government)
Responsible Party: Sponsor-Investigator, Chan-Sik Kim, Principal Investigator, Korea Institute of Oriental Medicine
Organization: Korea Institute of Oriental Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KIOM_2301_DED_USL
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard-dose USL group (Experimental): 2 tablets(1 USL, 1 placebo) b.i.d for 12 weeks
  Interventions: Drug: USL; Drug: USL Placebo
- High-dose USL group (Experimental): 2 tablets(2 USL) b.i.d for 12 weeks
  Interventions: Drug: USL
- Placebo group (Placebo Comparator): 2 tablets(2 placebo) b.i.d for 12 weeks
  Interventions: Drug: USL Placebo

INTERVENTIONS:
Drug: USL — 500mg of Achyranthis Radix Extract
  Arms: High-dose USL group; Standard-dose USL group
Drug: USL Placebo — USL Placebo
  Arms: Placebo group; Standard-dose USL group

SUMMARY:
The objective is to compare the USL and placebo in terms of efficacy and safety, and to determine the appropriate dosage.

DETAILED DESCRIPTION:
This study is a phase 2, dose-finding, double-blind, randomized placebo-controlled trial of two different doses of USL compared with placebo. A total of 120 patients, aged over 19 years, with Corneal staining score(Oxford grading) ≥ 2 or TBUT < 10 sec and OSDI ≥ 10 points will be recruited at Daejeon University Daejeon Korean Medicine Hospital. Patients will take medications two times daily for 12 weeks, with 5 visiting days(screening, week 0, week 6, week 12, week 14).

ELIGIBILITY:
Inclusion Criteria:

* Aged over 19
* Screening both eyes, the corrected visual acuity is 0.2 or more
* Subjects with Fluorescein Corneal Staining score (Oxford grading) ≥ 2 or TBUT test ≤10 at screening
* Subjects with OSDI ≥ 13
* Subjects who voluntarily agreed to participate in this clinical study in written form

Exclusion Criteria:

* Current or history of ocular disorders possibly affecting the study results (ocular surgery, trauma, diseases) as followings within 2 months:

  1. Abnormal eyelid function: disorders of the eyelids or eyelashes
  2. Ocular allergies or currently under the treatment of allergic diseases of the eye (topical ocular mast cell stabilizer, antihistamine use, etc.)
  3. Cicatricial keratoconjunctivitis caused by herpetic keratopathy, conjunctival scarring (alkali damage, Steven-Johnson syndrome, cicatricial pemphigoid), pterygium, pinguecula, lack of congenital lacrimal, neurogenic keratitis, keratoconus, corneal transplantation
* Those with acute eye inflammation/infection within 1 month
* Those who have undergone eye surgery (including LASIK/LASIK) within 3 months
* Those who had taken lacrimal punctal occlusion, cauterization of the punctum, or intense pulsed light procedure within 3 months
* Those who wear contact lenses within 72 hours of screening or plan to wear contact lens during the study period
* Intraocular pressure (IOP)> 25 mmHg in more than one side
* Autoimmune disease (e.g., Sjogren's syndrome, Rheumatoid arthritis, systemic lupus erythematosus, Graves' disease)
* Those who have used cyclosporine or diquafosol use in any form (systemic, topical) within 1 month
* Medical condition or history within 1 month to be treated with topical agents besides artificial tears (glaucoma, ocular allergy, ocular inflammation/infectious disease, etc.)
* Those who have taken or are taking steroid drugs or immunosuppressants (Azathioprine, Tacrolimus, Cyclosporin, Mycophenolate mofetil etc.) that may affect immune function within 3 months prior to screening
* Those who had taken antihypertensive drugs such as antihistamine and beta blockers, diuretics, antidepressants (especially tricyclic antidepressants, Parkinson's treatment drugs, etc.) that can worsen dry eye cannot participate in this study
* Severe abnormal liver function tests (Alanine transaminase (ALT) or Aspartate transaminase (AST) values ≥ 2 times the upper limit of normal) and abnormal renal function (Creatinine values ≥ 2 times the upper limit of normal)
* Genetic disorders, such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Comorbidities that may interrupt the treatment of cancers or clinically significant disorders of the kidney, liver, psychiatric system, cardiovascular system, respiratory system, endocrine system, and central nervous system, the safety assessment, or completion of this clinical study
* Unregulated hypertension (high blood pressure of 160 mmHg in the condenser or high blood pressure exceeding 100 mmHg in the relaxation period)
* Unregulated diabetes (fasting blood sugar (FBS) exceeding 180 mg/dL)
* Hepatitis A (active) or hepatitis B (active) or hepatitis C
* History of hypersensitivity reaction to active ingredients or excipients of the investigational product
* History of excessive alcohol use or drug addiction
* Pregnant or lactating women
* Those who did not agree to use contraception by medically permitted methods (e.g., surgical treatment of infertility, intrauterine device, condom or diaphragm, and injectable or insertable contraceptives) during the period from dosing of the investigational product to 90 days after the clinical study, among female subjects of childbearing potential and male subjects with the female partner
* Those who had experience of participating in a different clinical study within 4 weeks prior to participation in this clinical study
* Subjects who were determined to be ineligible to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TBUT(Tear break-up time) | Screening, 6 week, 12 week, 14 week
  The tear break-up time test measures the time in seconds. The time is from the last blinking to the point of tear layer defect or streak-like defect after blinking the eye with 1% of fluorescein.
  10 seconds or more as normal, between 5 and 10 seconds as mild dry eye syndrome, and 5 seconds or less as severe dry eye syndrome.

SECONDARY OUTCOMES:
OSDI(Ocular Surface Disease Index) | Screening, 6 week, 12 week, 14 week
  The Ocular Surface Disease Index consisted of 12 questions each of which included visual symptoms, visual work status, and environmental factors.
  The Ocular Surface Disease Index scores are ranged from 0 to 100, and the high score is the more severe the symptoms. The Ocular Surface Disease Index score is calculated as follows.
  : (Sum of all items answered × 25) / total number of questions answered
VAS(Visual analog scale) | 0 week, 6 week, 12 week, 14 week
  The Visual Analog Scale(VAS) score is 0 point for no symptom, 10 points for the most severe symptom, and the patient is asked to mark the degree of subjective pain symptoms as an integer.
Schirmer's test | 0 week, 6 week, 12 week, 14 week
  The eyes were wiped and the Schirmer test paper was inserted into the right eye at 1/3 of the lower eyelid without eye anesthesia and inserted into the left eye. After 5 minutes with the eyes closed, the Schirmer test paper was removed from the right side in the order of insertion and the left side removed. The wet length was measured in millimeters and the length of the midpoint was measured when the wet border was oblique.
Meibomian gland test | 0 week, 6 week, 12 week, 14 week
  By expression of eyelid, scoring of expressibility and quality of meibum will be tested. Form of secretion predominantly secreted by the eight meibomian glands in the center of the lid was evaluated as follows. grade 0, clear meibum is easily expressed; grade 1, cloudy meibum is expressed with mild pressure; grade 2, cloudy meibum is expressed with more than moderate pressure; and grade 3, meibum cannot be expressed even with the hard pressure. Higher score means a worst outcome.
Fluorescein corneal staining score - Oxford grading | Screening, 6 week, 12 week, 14 week
  The degree of corneal inflammation is scored (total of 5 points) according to the Oxford grading scale from 0 (no staining, A) to 5 (severe, confluent staining, >E).
SPEED-II (Standard Patient Evaluation for Eye Dryness-II) | 0 week, 6 week, 12 week, 14 week
  The SPEED questionnaire was designed in order to quickly track the progression of dry eye symptoms over time. This questionnaire gives a score from 0 to 28 that is the result of 8 items that assess frequency and severity of symptoms. The symptoms assessed include dryness, grittiness, scratchiness, irritation, burning, watering, soreness, and eye fatigue. The questionnaire further assesses whether these symptoms were not problematic, tolerable, uncomfortable, bothersome, or intolerable.
Biomarkers | 0 week, 12 week
  The levels of IL-1β, IFN-γ, TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Sik Kim, PhD, Principal Investigator — Korea Institute of Oriental Medicine

IPD SHARING:
Plan to Share IPD: No